CLINICAL TRIAL: NCT04502823
Title: Management of Fetal Growth Restriction at Term: Angiogenic Factors Versus Feto-placental Doppler (GRAFD Trial)
Brief Title: Management of Fetal Growth Restriction at Term: Angiogenic Factors Versus Feto-placental Doppler
Acronym: GRAFD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR(AMI)527/2019
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2021-07

CONDITIONS: Fetal Growth Retardation
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Clinical practice: Management by Doppler and CTG findings.
  In women allocated to the control group, the sFlt-1/PlGF result will be blinded to caregivers. Routine Doppler-based clinical care will be used to counsel women. Following the Doppler classification:
  * Fetuses with an EFW below the 3rd centile or below the 10th centile accompanied by any impaired fetoplacental Doppler, elective delivery will be recommended immediately (within 24h) at ≥37 weeks.
  * Fetuses with an EFW above the 3rd centile without any fetoplacental Doppler abnormality, elective delivery will be recommended at at ≥40 weeks.
- Intervention Group (Experimental): Management based on sFlt-1/PlGF values
  Interventions: Procedure: Management based on sFlt-1/PlGF values

INTERVENTIONS:
Procedure: Management based on sFlt-1/PlGF values — In women allocated to the intervention group, the sFlt-1/PlGF result will be revealed to the investigators that will act according to the results of sFlt/PlGF:
  * Fetuses with sFlt-1/PlGF ≥38, elective delivery will be recommended immediately (within 24h) at ≥37 weeks.
  * Fetuses with sFlt-1/PlGF <38 weekly follow up will be recommended and delivery at ≥40 weeks.
  Arms: Intervention Group

SUMMARY:
Open randomized non-inferiority controlled trial to examine the use of angiogenic factors (instead of feto-placental Doppler) for fetal growth restriction at term to reduce the rate of labor inductions, without worsening perinatal outcomes.

DETAILED DESCRIPTION:
Pregnant women with estimated fetal weight (EFW) < 10th centile between 36+0 and 37+6 weeks of gestation (WG) will receive complete ultrasonographic assessment consisting of feto-placental Doppler, amniotic fluid measurement and biophysical profile assessment. The cases not meeting any exclusion criteria will be offered to participate in this trial. After giving their informed consent a blood sample will be drawn in all of them and they will undergo randomization into two arms.

1. Intervention arm: In women allocated to the intervention group, the soluble fms-like tyrosine kinase/placental growth factor (sFlt-1/PlGF) result will be revealed to the investigators that will act according to the results of sFlt/PlGF:

   * Fetuses with sFlt-1/PlGF ≥38, elective delivery will be recommended at ≥37 weeks.
   * Fetuses with sFlt-1/PlGF <38, weekly follow up will be recommended until delivery (at ≥40 weeks).
2. Control arm: In women allocated to the control group, the sFlt-1/PlGF result will be blinded to caregivers. Routine Doppler-based clinical care will be used to counsel women. Following the Doppler classification:

   * Fetuses with EFW below the 3rd centile or below the 10th centile accompanied by any impaired fetoplacental Doppler, elective delivery will be recommended at at ≥37 weeks.
   * Fetuses with EFW above the 3rd centile without any fetoplacental Doppler abnormality, elective delivery will be recommended at at ≥40 weeks.

In both arms, fetuses will receive weekly follow-up from randomization to delivery consisting on feto-placental Doppler sFlt-1/PlGF and CTG. If any of the following is present at any time, earlier delivery will be recommended:

* sFlt-1/PlGF ≥38 (only in the intervention group),
* absent or reverse end-diastolic flow at the umbilical artery Doppler or DV PI>95th centile
* non-reassuring CTG
* preeclampsia
* diminished fetal movements
* biophysical profile ≤ 6 or oligohydramnios (deepest pocket <2 cm).

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women ≥ 16 years of age.
2. Singleton pregnancy.
3. Ultrasonographic estimated fetal weight <10th centile.
4. Gestational age between 36+0 and 37+6 weeks.

Exclusion Criteria:

1. Major fetal malformations or genetic disorders.
2. Fetal death.
3. Absent or reverse end-diastolic flow in umbilical artery Doppler or DV PI>95th centile.
4. Non-reassuring cardiotocography (CTG).
5. Preeclampsia.
6. Diminished fetal movements.
7. Biophysical profile ≤ 6.
8. Oligohydramnios
9. Refusal to give informed consent.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnant women
Enrollment: 1088 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2022-12-18 (Actual); Study Completion 2022-12-18 (Actual)

PRIMARY OUTCOMES:
Adverse perinatal outcomes | 4-6 weeks
  Cesarean delivery for non-reassuring fetal status or neonatal acidosis (artery cord potential of hydrogen (pH) <7.15 + base excess > -12 milliequivalent/L)

SECONDARY OUTCOMES:
Rate of elective delivery | 4-6 weeks
  Percentage of women that required an elective delivery
Rate of Cesarean delivery | 4-6 weeks
  Percentage of women that required a Cesarean delivery
Rate of Induction of labor | 4-6 weeks
  Percentage of women that required an induction of labor
Rate of neonatal admission in intensive care unit | 4-6 weeks
  Percentage of newborns that required admission in intensive care
Time of neonatal admission in intensive care unit | 4-6 weeks
  Days in in intensive care of newborns that required admission
Rate of preeclampsia | 4-6 weeks
  Percentage of women that developed preeclampsia
Rate of neonatal complications | 4-10 weeks
  Percentage of newborns with adverse outcomes (composite)
Rate of maternal complications | 4-6 weeks
  Percentage of women with adverse outcomes (composite)
Rate of perinatal complications | 4-6 weeks
  Percentage of perinatal adverse outcomes (composite)
Rate of total deliveries at <37, <38, <39 and <40 weeks of gestation | 4-6 weeks
  Percentage of women that delivered at <37, <38, <39 and <40 weeks of gestation
Rate of elective deliveries at <37, <38, <39 and <40 weeks of gestation | 4-6 weeks
  Percentage of women that delivered electively at <37, <38, <39 and <40 weeks of gestation
Rate of newborns with birthweight <2000 and <2500 grams | 4-6 weeks
  Percentage of women that delivered a newborn with a birthweight <2000 and <2500 grams

CONTACTS AND LOCATIONS:
Overall Officials: Manel Mendoza, PhD, Principal Investigator — Vall d'hebron Institut de Recerca
Locations (20):
- Spain (20):
  - Hospital Universitario de A Coruña, A Coruña
  - Hospital General de Alicante, Alicante
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitari Vall d'hebron, Barcelona
  - Hospital Universitario de Cabueñes, Cabueñes
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitario de Getafe, Getafe
  - Hospital Universitari Doctor Josep Trueta, Girona
  - Hospital Sant Joan de Deu de Manresa, Manresa
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Son Llàtzer, Palma de Mallorca
  - Consorci Corporació Sanitària Parc Taulí de Sabadell, Sabadell
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Universitari Joan XXIII, Tarragona
  - Hospital de Terrassa, Terrassa
  - Hospital Universitari Mútua Terrassa, Terrassa
  - Hospital Universitario de Torrejon, Torrejón de Ardoz
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza

REFERENCES:
- [Derived] Garcia-Manau P, Bonacina E, Martin-Alonso R, Martin L, Palacios A, Sanchez-Camps ML, Lesmes C, Hurtado I, Perez E, Tubau A, Ibanez P, Alcoz M, Valino N, Moreno E, Borrero C, Garcia E, Lopez-Quesada E, Diaz S, Broullon JR, Teixidor M, Chulilla C, Ferrer-Costa R, Gil MM, Lopez M, Ramos-Forner GM, Blanco JE, Moreno A, Lazaro-Rodriguez M, Vaquerizo O, Soriano B, Fabre M, Gomez-Valencia E, Cuina A, Alayon N, Sainz-Bueno JA, Vives A, Esteve E, Ocana V, Lopez MA, Maroto A, Carreras E, Mendoza M. Angiogenic factors versus fetomaternal Doppler for fetal growth restriction at term: an open-label, randomized controlled trial. Nat Med. 2025 Mar;31(3):1008-1015. doi: 10.1038/s41591-024-03421-9. Epub 2025 Jan 7. PMID 39775039
- [Derived] Garcia-Manau P, Mendoza M, Bonacina E, Martin-Alonso R, Martin L, Palacios A, Sanchez ML, Lesmes C, Hurtado I, Perez E, Tubau A, Ibanez P, Alcoz M, Valino N, Moreno E, Borrero C, Garcia E, Lopez-Quesada E, Diaz S, Broullon JR, Teixidor M, Chulilla C, Gil MM, Lopez M, Candela-Hidalgo A, Salinas-Amoros A, Moreno A, Morra F, Vaquerizo O, Soriano B, Fabre M, Gomez-Valencia E, Cuina A, Alayon N, Sainz JA, Vives A, Esteve E, Ocana V, Lopez MA, Maroto A, Carreras E. The Fetal Growth Restriction at Term Managed by Angiogenic Factors Versus Feto-Maternal Doppler (GRAFD) Trial to Avoid Adverse Perinatal Outcomes: Protocol for a Multicenter, Open-Label, Randomized Controlled Trial. JMIR Res Protoc. 2022 Oct 11;11(10):e37452. doi: 10.2196/37452. PMID 36222789